CLINICAL TRIAL: NCT00580879
Title: Does Antenatal Fetal Head Circumference Predict Anal Sphincter Injury, a Prospective Study
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Karen Noblett, Associate Professor, University of California, Irvine Medical Center
Other Study IDs: 2005-4575
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Anorectal Sphincter Laceration; Pelvic Floor Dysfunction
Keywords: Anorectal sphincter laceration; Pelvic floor dysfunction; Sphincter tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to see if fetal head circumference can be used as a predictor for who will experience a sphincter laceration while delivering.

DETAILED DESCRIPTION:
Even though much work has been invested in trying to identify risk factors that can predict which population will suffer from sphincter tears and other pelvic floor trauma, the epidemiology is still poorly understood. Factors that have been implicated to include operative vaginal delivery, birth weight, and primaparity. Up to this point little focus has been placed on antenatal factors that would help predict and prevent sphincter disruptions. At the time of birth the infant's head is the largest part of the body. Thus, head circumference of the infant may be able to predict which subjects is more likely to suffer from sphincter disruption. Thus, this study aims to determine whether or not fetal head circumference measured antenatally is predictive of pelvic floor trauma.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous subjects at least 18 years of age
* Gestational age greater than or equal to 36 weeks and upto 42 weeks gestation
* Subjects must have give written informed consent to participate in this study
* Subjects must be planning to deliver at UCI

Exclusion Criteria:

* Subjects less than 18 years of age
* Subjects with a previous delivery
* Subjects with previous colorectal surgery or hemorrhoidal surgery
* Subjects with a history of irritable bowel syndrome, ulcerative colitis, or Crohn's disease
* Subjects with a history of colon or rectal cancer
* Gestational age less than 36 weeks
* Cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in 36 weeks and upto 42 weeks of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Fetal head circumference and position, maternal pelvis, infant weight, maternal weight, length of the second stage, the incidence of sphincter tears as diagnosed by transvaginal ultrasound as well as the incidence of fecal urgency and incontinence. | 6 Months

SECONDARY OUTCOMES:
The magnitude of the effect of other factors such as maternal obesity, maternal age, duration of labor and pelvimetry on the risk of anorectal lacerations will be examined. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Noblett, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States